CLINICAL TRIAL: NCT02995902
Title: FLT-PET/DW-MRI for Detection of Brain Metastases and Early Therapy Evaluation in Patients With Small Cell Lung Cancer
Acronym: SIBES II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tine Nøhr Christensen, MD, research fellow, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 307_14
Record Dates: First submitted 2016-12-09; First posted 2016-12-19 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

ARMS (1):
- FLT-PET/MRI (Experimental)
  Interventions: Device: FLT-PET; Device: MRI

INTERVENTIONS:
Device: FLT-PET
Device: MRI

SUMMARY:
The purpose of the study is to determine the value of FLT-PET early after initiated chemotherapy in patients with small cell lung cancer, and to determine whether MRI of the brain should be performed routinely in these patients.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven small cell lung cancer
* referred for standard chemotherapy
* oral and written informed consent

Exclusion Criteria:

* metal or electronical devices in the body not compatible with MRI of brain or thorax
* pregnancy or lactation
* communication difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year
Disease free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, MD phD MDSci, Study Chair — Dept of Clinical Physiology, Nuclear medicine and PET, Rigshospitalet, Denmark
Locations (1):
- Dept. of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Result] Christensen TN, Langer SW, Villumsen KE, Johannesen HH, Lofgren J, Keller SH, Hansen AE, Kjaer A, Fischer BM. 18F-fluorothymidine (FLT)-PET and diffusion-weighted MRI for early response evaluation in patients with small cell lung cancer: a pilot study. Eur J Hybrid Imaging. 2020 Jan 27;4(1):2. doi: 10.1186/s41824-019-0071-5. PMID 34191195